CLINICAL TRIAL: NCT00491517
Title: Sirolimus Treatment in Patients With ADPKD
Brief Title: Sirolimus Treatment in Patients With Autosomal Dominant Polycystic Kidney Disease: Renal Efficacy and Safety
Acronym: SIRENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIRENA; 2006-003427-37 (EudraCT Number)
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental)
  Interventions: Drug: Sirolimus
- conventional therapy (Active Comparator)
  Interventions: Drug: conventional therapy

INTERVENTIONS:
Drug: Sirolimus — Patients will be given Sirolimus starting at the oral daily dose of 3 mg with periodically whole blood level measurements. The daily dose will be adjusted to keep sirolimus concentration within 10-15 ng/ml.
  Arms: Sirolimus
Drug: conventional therapy — Antihypertensive drugs for patients with high blood pressure.
  Arms: conventional therapy

SUMMARY:
Autosomal-Dominant Polycystic Kidney Disease (ADPKD) is the most common hereditary renal disease, characterized by the progressive development of fluid-filled cysts in the kidney leading to progressive loss of renal function and eventually to renal failure. It is responsible for 8% to 10% of the cases of end stage renal disease (ESRD) in Western countries. ADPKD progression is largely dependent on the development and growth of the cysts and secondary disruption of the normal tissue. Renoprotective interventions in ADPKD - in addition to achieve maximal reduction of arterial blood pressure and proteinuria and to limit the effects of additional potential promoters of disease progression such as dyslipidemia, chronic hyperglycemia or smoking - should also be specifically aimed to correct the dysregulation of epithelial cell growth, secretion, and matrix interactions characteristic of the disease. Genetically in the ADPKD three different genes are implicated (PKD1 85% of the cases, PKD2 15% and probably PDK3 not yet identified). PKD1 gene encodes a protein named polycystin-1 (PC1). Defect in PC1 lead to aberrant activation of the enzyme mTOR in the epithelial cells of the renal tubules which eventually leads to abnormal proliferation of these cells and cysts generation.

Sirolimus (Rapamycin) is an immunosuppressant mostly used for the management of kidney transplant recipients. This drug by very specifically and effectively inhibiting mTOR, exerts antiproliferative and growth inhibiting effects and could be extremely important for the inhibition of cyst progression in ADPKD. Animal models of ADPKD have shown that short-term treatment with sirolimus resulted in dramatic reduction of kidney size, prevented the loss of kidney function, and lowered cyst volume density. Similarly, retrospective observations from kidney transplant recipients have documented that sirolimus treatment reduced kidney volumes by 25%, whereas there was no effect in patients not given the drug.

Overall, these findings provide the basis for designing a prospective study in ADPKD patients aimed to document the efficacy of sirolimus treatment in preventing further increase or even reducing the total kidney volume and the renal volume taken up by small cysts, eventually halting kidney disease progression. It is a 6 month treatment with sirolimus compared to conventional therapy in adult patients with ADPKD and normal renal function or mild to moderate renal insufficiency.

DETAILED DESCRIPTION:
Introduction Autosomal-Dominant Polycystic Kidney Disease (ADPKD) is the most common hereditary renal disease, responsible for 8% to 10% of the cases of end stage renal disease (ESRD) in Western countries. The disease is characterized by the progressive development of fluid-filled cysts in the kidney. The renal cysts originate from the epithelia of the nephrons and are lined by a single layer of cells that have a higher rate of cellular growth and proliferation. At comparable levels of blood pressure control and proteinuria, patients with ADPKD have faster decline in glomerular filtration rate (GFR) than those with other renal diseases and do not seem to benefit to the same extent of ACE inhibitor therapy. Thus, renoprotective interventions in ADPKD - in addition to achieve maximal reduction of arterial blood pressure and proteinuria and to limit the effects of additional potential promoters of disease progression such as dyslipidemia, chronic hyperglycemia or smoking - should also be specifically aimed to correct the dysregulation of epithelial cell growth, secretion, and matrix interactions characteristic of the disease.

ADPKD shows genetic heterogeneity, with at least three different genes implicated: the PKD1 gene (85% of the cases), the PKD2 (15% of the cases), and probably a PDK3 gene (not yet identified). PKD1 gene was identified more than a decade ago, the development of treatment strategies has been hampered by a lack of understanding of the function of polycystin-1 (PC1), the protein encoded by the PKD1 gene. However, a new function of PC1 has been recently identified, which suggests a possibility for future treatment options. Indeed, it has been reported that PC1 tail interacts with tuberin, the product of the TSC2 gene. The main function of tuberin is to inactivate the Ser/Thr kinase mTOR which, in turn, promotes phosphorylation of two proteins, S6-kinase and 4E-BP1. mTOR activity has been linked to increased cell growth, proliferation, apoptosis and changes in differentiation. Researchers have subsequently shown that in ADPKD experimental animal models cyst lining epithelial cells exhibited very high mTOR activity, and hypothesized that PC1 normally suppresses mTOR activity and that defects in PC1 (and in other proteins) lead to aberrant mTOR activation. Of interest, all these proteins are localized to primary cilia or renal epithelial cells or to the basal bodies from which cilia emanate. This finding has led to the view that loss of cilia function leads to cysts formation in the kidney. The finding that mTOR is inappropriately activated in polycystic kidney disease mouse models suggests that mTOR activation may be a consequence of the loss of cilia function. If mTOR is such a converging point, it would be worthwhile as possible drug target for treatment of renal cystic disorders.

Sirolimus is an immunosuppressant mostly used for the management of kidney transplant recipients. This drug by very specifically and effectively inhibiting mTOR, exerts antiproliferative and growth inhibiting effects that might serve preventing uncontrolled tubular cell proliferation and could be extremely important for the inhibition of cyst progression in APKD. Interestingly, studies in rat models of ADPKD have shown that short-term treatment with sirolimus resulted in dramatic reduction of kidney size, prevented the loss of kidney function, and lowered cyst volume density. Similarly, retrospective observations from kidney transplant recipients have documented that sirolimus treatment reduced kidney volumes by 25%, whereas there was no effect in patients not given the drug.

Overall, these findings provide the basis for designing a prospective study in ADPKD patients aimed to document the efficacy of sirolimus treatment in preventing further increase or even reducing the total kidney volume and the renal volume taken up by small cysts, eventually halting kidney disease progression. As an additional aim of the present study, we will assess the safety profile of sirolimus, when given to ADPKD patients.

Aim The general aim of this study is to assess the efficacy and safety of 6 month treatment with sirolimus (on the top of the best available therapy) as compared to conventional therapy in adult patients with ADPKD and normal renal function or mild to moderate renal insufficiency. In particular we will compare the change over baseline of the total kidney volume volume in sirolimus and conventional treatment ADPKD groups during 6 month follow-up.

Study Design This will be a randomized, longitudinal, open, cross-over study with a baseline evaluation and 6 month treatment period with sirolimus given in addition to conventional anti-hypertensive therapy to appropriately control blood pressure, in ADPKD patients (n=16).

Sirolimus Patients will be given sirolimus starting at the oral daily dose of 3 mg, with periodical whole blood level measurements. The daily dose will be adjusted to keep sirolimus concentration within 10-15 ng/ml. Drug levels will be assessed at day 5 after starting treatment and every two weeks for the first month; subsequently sirolimus concentrations will be monitored at monthly intervals (or 5 days after drug dose adjustments) until the end of the study.

Conventional Therapy There is no specific therapy for ADPKD patients. Conventional treatment relates usually to the administration of antihypertensive drugs for patients with high blood pressure. Thus, for the present study, no major change in antihypertensive treatment should be introduced throughout the whole study period unless deemed clinically necessary (the reason of the changes should be, however, clearly explained in the CRF). Only small changes in the doses of the ongoing treatments are recommended in order to maintain the same level of blood pressure control (target systolic/diastolic blood pressure <130/80 mnHg). This approach is aimed to minimize the confounding effect of any change in concomitant treatments on some efficacy variables (such as urinary protein excretion rate).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinical and ultrasound diagnosis of ADPKD
* GFR >40 ml/min/1.73 m2 (estimated by the 4 variable MDRD equation)
* Urinary protein excretion rate ≤ 0.5 g/ 24 hrs
* Written informed consent

Exclusion Criteria:

* Diabetes
* Urinary protein excretion rate >0.5 g/ 24 hrs or abnormal urinalysis suggestive of concomitant, clinically significant glomerular disease
* Urinary tract lithiasis, infection or obstruction
* Cancer
* Psychiatric disorders and any condition that might prevent full comprehension of the purposes and risks of the study
* Pregnancy, lactation or child bearing potential and ineffective contraception (estrogen therapy in post menopausal women should not be stopped)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-03; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Total kidney volume (estimated by computed tomography, CT) in sirolimus and conventional treatment ADPKD groups during 6 month follow-up. | At 0,6 and 12 months.

SECONDARY OUTCOMES:
Renal cyst volume, renal parenchymal volume and renal intermediate volume. | At 0,6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (1):
- Hospital "Azienda Ospedaliera Ospedali Riuniti di Bergamo" Unit of Neprology and Dialysis, Bergamo, Italy

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039